CLINICAL TRIAL: NCT06564519
Title: Check Yourself Before You Wreck Yourself: A Wearable Biofeedback Device to Decrease Surgical Resident's Time in a Non-upright Posture and Work-related Musculoskeletal Pain
Brief Title: Resident Posture Biofeedback Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00115419
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Postural; Strain; Healthy
Keywords: Biofeedback; Surgery; Surgical Resident
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Residents (Other): This is a single arm study. All Resident participants will use the posture biofeedback device.
  Interventions: Device: Posture Biofeedback Device

INTERVENTIONS:
Device: Posture Biofeedback Device — Participants will wear a commercially available posture training device for a two-week tracking period and a two-week training period while performing laparoscopic procedures.

SUMMARY:
While a majority of surgical ergonomic studies have been evaluating attending surgeons, few have evaluated surgical ergonomics within the surgical resident. Biofeedback devices can be partnered with education and geared towards surgical residents to decrease current and future musculoskeletal disorders, which may in turn lead to longer and more fulfilling careers.

DETAILED DESCRIPTION:
This study aims to use a commercially-available posture training device for surgical residents that sends biofeedback in the form of a gentle vibration if posture has deviated from the upright (neutral) position for a long period of time. For residents performing minimally-invasive procedures with a laparoscopic approach, our overarching hypothesis is that the time spent in a non-upright position will be less after using the posture biofeedback device compared with before. The study hypothesizes that residents will report fewer complaints related to musculoskeletal pain after wearing the posture training device.

Residents completing general surgery rotations will be recruited and wear a biofeedback device for about four weeks while performing laparoscopic procedures. Posture data from the device and survey data in the form of the Cornell Musculoskeletal Discomfort Questionnaire (CMDQ) will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Surgical residents with surgical experience of at least one year (Postgraduate year 2-5)
* Completing a one-month rotation at the study sites within the general surgery department during the study period

Exclusion Criteria:

* Clinically diagnosed inflammatory musculoskeletal disorders per self-report
* History of orthopedic surgery in the last six months per self-report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-11-02 (Actual); Study Completion 2025-11-02 (Actual)

PRIMARY OUTCOMES:
Time spent in upright vs non-upright position | week 1 to week 4]
  proportion (percentage) of time (minutes) in the upright position relative to the non-upright position during laparoscopic procedures

SECONDARY OUTCOMES:
Change in Self-reported musculoskeletal pain score | baseline to week 4
  Complaints related to musculoskeletal pain assessed using the Cornell Musculoskeletal Discomfort Questionnaire (CMDQ) - measures self-reported musculoskeletal discomfort for all body segments. 1 = low (score 1-2) 2 = moderate (score 3-4) 3 = high (score 5-7) 4 = very high (score 8-10 - higher scores meaning more discomfort

CONTACTS AND LOCATIONS:
Overall Officials: William Sherrill, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-08-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT06564519/ICF_000.pdf